CLINICAL TRIAL: NCT04964388
Title: Effect of GLP-1 Receptor Agonists on Trabecular Bone Score and Visceral Adiposity in Postmenopausal Women With Type 2 Diabetes Mellitus.
Brief Title: Effect of GLP-1 Receptor Agonists on Trabecular Bone Score
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Not able to recruit participants
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMississippi
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Results first posted 2024-07-24 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Osteoporosis, Postmenopausal; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- GLP-1 cohort (Experimental): Participants on GLP-1 receptor agonists
  Interventions: Drug: GLP-1 receptor agonist
- Non GLP-1 cohort (No Intervention): Participants not on GLP-1 receptor agonists

INTERVENTIONS:
Drug: GLP-1 receptor agonist — Diabetes medication
  Arms: GLP-1 cohort

SUMMARY:
This study will help determine the effect of Glucagon Like Peptide-1 (GLP-1)receptor agonists on bone strength in postmenopausal women with type 2 diabetes mellitus (T2DM)

DETAILED DESCRIPTION:
Postmenopausal women with diabetes mellitus have a higher risk of osteoporotic fractures, with significant associated mortality and morbidity. Osteoporosis is underdiagnosed in diabetes, as the bone mineral density (BMD) as currently measured is often normal despite underlying abnormalities. The trabecular bone score (TBS) is a novel modality to assess bone microarchitecture and accurately assess fracture risk in patients with diabetes. Due to increased co-prevalence of osteoporosis and diabetes mellitus, the potential effects of antidiabetic medications on fracture risk assume importance.

Based on findings in animal studies, we hypothesize that GLP-1 receptor agonists increase TBS in postmenopausal women with (T2DM). The investigators propose a prospective non-randomized study by enrolling 48 patients (24 in the GLP-1 group and 24 in the non-GLP group). Dual-energy X-ray Absorptiometry (DXA )scans, markers of bone formation, and resorption, and selected inflammatory markers will be assessed at baseline, six months, and one year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 Diabetes Mellitus
* Postmenopausal female
* Age >55 years
* Hemoglobin A1c between 7-10% within 6 months of the first visit.

Exclusion Criteria:

* Patients with type 1 Diabetes mellitus
* Patients with a history of GLP-1 receptor agonist/DPP4 inhibitor use
* eGFR <30 ml/min in the last 3 months
* Patients with a history of pancreatitis
* Personal or family history of medullary thyroid cancer
* Patients with a history of treatment with anti-osteoporosis agents
* Documented secondary osteoporosis
* Documented presence of prosthesis or devices in the spine
* Unwilling or unable to consent

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vishnu V Garla, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No
No sharing

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GLP-1 Cohort | Non GLP-1 Cohort
Started | 3 | 2
Completed | 0 | 0
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GLP-1 Cohort | Non GLP-1 Cohort | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 0 | 1 | 1
Age, Continuous [Median (Full Range); unit: years] | 58 [52 to 61] | 60 [54 to 67] | 58 [52 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Trabecular Bone Score
Description: The change in TBS from baseline to six months and one year after the initiation of a GLP-1 receptor agonist. TBS will be assessed by DXA scans done at baseline, six months and one year.
Time Frame: 12 months after index date
Population: Unfortunately at the time of enrollment the dexa scan was not functioning, after the machine was fixed we tried several times to contact the participants but could not get in touch with them. Therefore no dexa scans were done on the participants so no data was captured.
Arm/Group | GLP-1 Cohort | Non GLP-1 Cohort
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Inflammatory Markers and Bone Resorption Markers
Description: The change in inflammatory markers (IL-1, IL-6 and TNF-alpha) and bone resorption markers (C-telopeptide) at 6 and 12 months after starting GLP-1 receptor agonists as compared to baseline.
Time Frame: 12 months after index date
Population: Despite several attempts to get in touch with participants we could not get in touch with them therefore no data to report.
Arm/Group | GLP-1 Cohort | Non GLP-1 Cohort
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Visceral Fat Mass
Description: The change in visceral fat mass (measured by DXA) at 6 and 1 year after starting GLP-1 receptor agonists as compared to baseline.
Time Frame: 12 months after index date
Population: as for outcome 2
Arm/Group | GLP-1 Cohort | Non GLP-1 Cohort
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Sclerostin and Bone Formation Markers
Description: The change in levels of sclerostin, osteocalcin, and P1NP (as measured by commercial assays) from baseline to six months and one year after starting GLP-1 receptor agonist.
Time Frame: 12 months after index date
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The specific period of time over which each participant was assessed would have been one year However, none of the participants were lost to follow-up, so adverse events could not be assessed.
Arm/Group | GLP-1 Cohort | Non GLP-1 Cohort
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/88/NCT04964388/Prot_SAP_000.pdf